CLINICAL TRIAL: NCT00574106
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation for Cancer Treatment
Brief Title: A Study to Evaluate the Effect of Far Infrared Radiation for Cancer Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina, The Centre for Incurable Diseases, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-CAN-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Neoplasms
Keywords: Cancer; Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Infrared Radiation
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength)

SUMMARY:
Cancer is the number one killer in Canada and in most countries of the world. The investigators' initial assessment indicates that far infrared radiation has the potential to cure cancer.

DETAILED DESCRIPTION:
The investigators have identified a combination of methods for possible cancer treatment as follows:

1. Energy specific far infrared radiation (5 μm to 20 μm ). No x-rays, gamma rays etc. are used.
2. Oxygenation of the body cells
3. pH balance
4. Lifestyle changes, or
5. A combination of chemotherapy and (1), (2), (3) and (4) above.

ELIGIBILITY:
Inclusion Criteria:

* All cancer patients

Exclusion Criteria:

* non-cancer patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The effect of far infrared radiation on cancerous tumours | 1 year

SECONDARY OUTCOMES:
The effect on far infrared treatment on different kinds of cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada